CLINICAL TRIAL: NCT01190553
Title: Maintenance Therapy of Intravenous Amantadine in Patients With Idiopathic Parkinson Disease Who Are Not Optimally Treated With Anti Parkinson Medications
Brief Title: Pilot Study of Maintenance Therapy With Intravenous AMANTADINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Prof. Ruth Djaldetti, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0166-10-RMC
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-08

CONDITIONS: Parkinson Disease
Keywords: amantadine; parkinson disease; dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): IV amantadine treatment
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — Initiation: IV amantadine 200mg/500ml * 1/d for 3 days Maintenance: IV amantadine 200mg/500ml once per 6 weeks for 6 months
  Other Names: PK-Merz

SUMMARY:
This is a pilot study for Maintenance Intravenous Treatment with AMANTADINE in patient with PARKINSON'S Disease who are not well balanced with medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson disease
* Age<80
* Patients with no motor improvement under optimal treatment with anti parkinson medications
* Patients with moderate to severe dyskinesias
* Patients with PD with side effects who can not tolerate anti parkinson medications

Exclusion Criteria:

* Age>80
* Patients with Parkinson syndromes, vascular parkinsonism or drug-induced parkinsonism
* Patients with PD who developed adverse reactions to oral amantadine
* Contraindication of amantadine treatment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of UPDRS scores after 6 months of treatment | 6 months
Improvement of dyskinesias score. | 6 months